CLINICAL TRIAL: NCT07015255
Title: Assessing the Burden of Respiratory Syncytial Virus (RSV): the Assessment of the Burden of Respiratory Syncytial Virus (RSV) Across Different Age Groups and Risk Factors
Brief Title: Assessing the Burden of Respiratory Syncytial Virus (RSV)
Status: Not yet recruiting | Type: Observational
Sponsor: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Sponsor
Other Study IDs: DOH/ADHRTC/2025/361
Record Dates: First submitted 2025-05-16; First posted 2025-06-11 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Syncytial Virus (RSV) Infection; Acute Lower Respiratory Tract Infections; Bronchiolitis; Pneumonia; Chronic Respiratory Conditions
Keywords: Respiratory Syncytial Virus; RSV; RSV Infection; RSV in Infants; RSV in Adults; RSV Hospitalization; RSV Epidemiology; RSV Burden; RSV Risk Factors; Retrospective Study; Observational Study; ICU Admissions; RSV Mortality; RSV Cost Analysis; RSV Complications; Asthma and RSV; Bronchiolitis; Pneumonia; Recurrent Wheezing; RSV Surveillance; RSV-Related Comorbidities
MeSH Terms: conditions — Infections; Bronchiolitis; Pneumonia; Respiratory Syncytial Virus Infections; Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infants, adults, elderly, and high-risk patients with confirmed RSV infection (2018-2024).: This retrospective study includes patients of all ages with confirmed Respiratory Syncytial Virus (RSV) infection from January 2018 to December 2024, categorized into four cohorts: (1) Infants and young children, including those with risk factors such as prematurity, low birth weight, and chronic lung or heart disease; (2) Adults aged 18-64 years with or without comorbidities; (3) Elderly adults aged 65 and older, with focus on severe outcomes and mortality; and (4) High-risk individuals across all age groups with underlying conditions such as asthma, COPD, diabetes, immunosuppression, Down syndrome, or cystic fibrosis. No interventions are administered; the study analyzes existing data to assess RSV burden, ICU admissions, long-term health impacts, and associated healthcare costs.

SUMMARY:
This study examines the impact of Respiratory Syncytial Virus (RSV) on people of all ages, from infants to the elderly. It uses hospital records collected between January 2018 and December 2024 to understand:

* How often does RSV occur
* Who is most at risk
* The long-term and financial effects of RSV

DETAILED DESCRIPTION:
This study is designed to analyze the impact of Respiratory Syncytial Virus (RSV) across different age groups. It focuses on how often RSV occurs, who is most at risk, and its long-term and financial effects. The study uses existing hospital records from SEHA facilities between January 2018 and December 2024. This is a retrospective observational study, meaning no new tests or treatments are given. Researchers look at medical records from past patients who were diagnosed with RSV. Anonymized data is collected from SEHA's Electronic Medical Records (EMR) and laboratory systems. Only patients with confirmed RSV infections are included.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with a confirmed diagnosis of RSV infection
* Patients admitted to a SEHA hospital or healthcare facility between January 2018 and December 2024
* Patients with documented data in the SEHA electronic medical record (EMR) system

Exclusion Criteria:

* Patients with suspected RSV infection that is not laboratory-confirmed
* Patients without sufficient data in the SEHA EMR system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes all patients of any age who have a laboratory-confirmed diagnosis of Respiratory Syncytial Virus (RSV) infection recorded in the SEHA electronic medical records between January 2018 and December 2024. The population spans from newborn infants to elderly adults, including those with underlying medical conditions such as chronic lung disease, heart disease, immunosuppression, and other comorbidities that may influence RSV severity. Both hospitalized patients and those diagnosed in outpatient settings within SEHA healthcare facilities are included. The study aims to represent the full spectrum of RSV disease burden, clinical outcomes, risk factors, long-term health impacts, and healthcare costs across diverse demographic groups in the UAE.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Burden of RSV Infection Across All Age Groups | January 2018 - December 2024
  Measurement of the incidence of confirmed RSV infections in patients of all ages using SEHA hospital data from January 2018 to December 2024.
Burden of RSV Infection Across All Age Groups | January 2018 - December 2024
  Measurement of the prevalence of confirmed RSV infections in patients of all ages using SEHA hospital data from January 2018 to December 2024.

SECONDARY OUTCOMES:
Identification of Risk Factors for Severe RSV Infection | January 2018 - December 2024
  Analysis of clinical, demographic, and comorbidity data to identify key risk factors associated with severe RSV infection outcomes.
Proportion of Hospital Admissions Due to RSV | January 2018 - December 2024
  Evaluation of the percentage of total hospital admissions attributed to RSV infections.
ICU Admission Rates for RSV-Infected Patients | January 2018 - December 2024
  Measurement of the proportion of RSV patients requiring ICU care.
Financial Burden of RSV Infection | January 2018 - December 2024
  Assessment of direct medical costs associated with RSV hospitalization and ICU care.
Incidence of Recurrent Wheezing and Asthma Diagnosis Following RSV Infection | Up to 12 months post-infection
  Evaluation of long-term respiratory complications, specifically:
  1. Clinically diagnosed asthma using standardized clinical criteria (e.g., based on ICD-10 codes or physician diagnosis recorded in medical records)
  2. Recurrent wheezing episodes, defined as ≥3 wheezing episodes confirmed by clinical examination or parent report within 12 months post-infection, assessed via structured caregiver questionnaires and medical record review.
RSV-Associated Mortality Rates | January 2018 - December 2024
  Analysis of death rates among RSV-positive patients, including 30-day mortality post-admission.
Long-Term Respiratory Outcomes Following RSV Infection | Up to 12 months post-infection
  Evaluation of post-RSV respiratory complications such as asthma and recurrent wheezing.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Eldin Hussein, MD, Study Director — Abu Dhabi Health Services Company-SEHA; Nawal Alkaabi, MD, Principal Investigator — Abu Dhabi Health Services Company-SEHA
Locations (1):
- Sheikh Khalifa Medical City (Abu Dhabi Health Research Centre), SEHA, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felton DA. A time of 'firsts'. J Prosthodont. 2004 Mar;13(1):1-2. doi: 10.1111/j.1532-849X.2004.04011.x. No abstract available. PMID 15032890
- [Background] Zhou H, Thompson WW, Viboud CG, Ringholz CM, Cheng PY, Steiner C, Abedi GR, Anderson LJ, Brammer L, Shay DK. Hospitalizations associated with influenza and respiratory syncytial virus in the United States, 1993-2008. Clin Infect Dis. 2012 May;54(10):1427-36. doi: 10.1093/cid/cis211. Epub 2012 Apr 10. PMID 22495079
- [Background] Hall CB, Weinberg GA, Iwane MK, Blumkin AK, Edwards KM, Staat MA, Auinger P, Griffin MR, Poehling KA, Erdman D, Grijalva CG, Zhu Y, Szilagyi P. The burden of respiratory syncytial virus infection in young children. N Engl J Med. 2009 Feb 5;360(6):588-98. doi: 10.1056/NEJMoa0804877. PMID 19196675
- [Background] Wassmer SC, Lepolard C, Traore B, Pouvelle B, Gysin J, Grau GE. Platelets reorient Plasmodium falciparum-infected erythrocyte cytoadhesion to activated endothelial cells. J Infect Dis. 2004 Jan 15;189(2):180-9. doi: 10.1086/380761. Epub 2004 Jan 9. PMID 14722881
- [Background] Callen A, Diener-West M, Zeitlin PL, Rubenstein RC. A simplified cyclic adenosine monophosphate-mediated sweat rate test for quantitative measure of cystic fibrosis transmembrane regulator (CFTR) function. J Pediatr. 2000 Dec;137(6):849-55. doi: 10.1067/mpd.2000.109198. PMID 11113843
- [Background] Falsey AR, Hennessey PA, Formica MA, Cox C, Walsh EE. Respiratory syncytial virus infection in elderly and high-risk adults. N Engl J Med. 2005 Apr 28;352(17):1749-59. doi: 10.1056/NEJMoa043951. PMID 15858184
- [Background] Joury J, Al Kaabi N, Al Dallal S, Mahboub B, Zayed M, Abdelaziz M, Onwumeh-Okwundu J, Fletcher MA, Kumaresan S, Ramachandrachar BC, Farghaly M. Retrospective Analysis of RSV Infection in Pediatric Patients: Epidemiology, Comorbidities, Treatment, and Costs in Dubai (2014-2023). J Health Econ Outcomes Res. 2024 Nov 5;11(2):133-144. doi: 10.36469/001c.123889. eCollection 2024. PMID 39575134
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- See also: World Health Organization (WHO) - RSV Fact Sheet — https://www.who.int/news-room/fact-sheets/detail/respiratory-syncytial-virus-(rsv)
- See also: Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. — https://pubmed.ncbi.nlm.nih.gov/20399493/
- See also: Respiratory syncytial virus infection in elderly and high-risk adults. — https://pubmed.ncbi.nlm.nih.gov/15858184/
- See also: Rates of hospitalization for respiratory syncytial virus infection among children in Medicaid. — https://pubmed.ncbi.nlm.nih.gov/11113843/
- See also: Updated guidance for palivizumab prophylaxis among infants and young children at increased risk of hospitalization for respiratory syncytial virus infection. — https://doi.org/10.1542/peds.2014-1665
- See also: Risk factors for severe respiratory syncytial virus infection in elderly persons. — https://pubmed.ncbi.nlm.nih.gov/14722881/
- See also: The burden of respiratory syncytial virus infection in young children. — https://pubmed.ncbi.nlm.nih.gov/19196675/
- See also: Hospitalizations associated with influenza and respiratory syncytial virus in the United States, 1993-2008. — https://pubmed.ncbi.nlm.nih.gov/22495079/
- See also: Economic impact of respiratory syncytial virus-related illness in the US: an analysis of national databases. — https://pubmed.ncbi.nlm.nih.gov/15032890/